CLINICAL TRIAL: NCT06625528
Title: The Efficacy of Lyophilized Platelet-Rich Fibrin in Treatment of Periodontal Intra-Bony Defects (A Comparative Clinical, Radiographic and Biochemical Study)
Brief Title: The Present Study Was Performed to Evaluate the Efficacy of Lyophilized-PRF in Treatment of Periodontal Intra-bony Defects
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa El-Dein Mohamed Maamoun Salatein, assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: periodontal treatments
Record Dates: First submitted 2024-09-26; First posted 2024-10-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Treatment of Periodontal Intra-bony Defects
Keywords: periodontitis; lyophilized-PRF; Periodontal intra-Bony Defects; Periodontal angular bone defect
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: The patients selected in this study will be randomly divided into 3 groups:
  Group I: Periodontitis patients with an intra-bony defect will be treated by open flap debridement.
  Group II: Periodontitis patients with an intra-bony defect will be treated by open flap debridement combined with the application of lyophilized platelet-rich fibrin.
  Group III: Periodontitis patients with an intra-bony defect will be treated by open flap debridement and lyophilized platelet-rich fibrin combined with nanocrystalline hydroxyapatite bone substitute.
  All patients will be evaluated clinically, radiographically and biochemically
Who Masked: Outcomes Assessor
Masking Description: The statistician and the evaluator were blinded, but the operator was not because of the nature of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- open flap debridement (Placebo Comparator): Immediately before surgery, patients rinsed with 0.12% chlorhexidine digluconate and povidone iodine solution was used to perform extra-oral antisepsis. The surgical site was anaesthetized. A mucoperiosteal flap was elevated and reflected followed by thorough debridement of all inflammatory granulation tissue from IBD until a sound, healthy bone surface was obtained. Root surface debridement was also performed. Copious irrigation with normal saline solution. The flap was repositioned and sutured.
  Interventions: Biological: open flap debridement
- lyophilized platelet rich fibrin (Active Comparator): Immediately before surgery, patients rinsed with 0.12% chlorhexidine digluconate and povidone iodine solution was used to perform extra-oral antisepsis. The surgical site was anaesthetized. A mucoperiosteal flap was elevated and reflected followed by thorough debridement of all inflammatory granulation tissue from IBD until a sound, healthy bone surface was obtained. Root surface debridement was also performed. Copious irrigation with normal saline solution. The lyophilized-PRF granules was hydrated with a few drops of normal saline then, it was applied and packed to fill defect. The flap was repositioned and sutured.
  Interventions: Biological: open flap debridement
- lyo-PRF and nanocrystalline hydroxyapatite bone graft (Active Comparator): Immediately before surgery, patients rinsed with 0.12% chlorhexidine digluconate and povidone iodine solution was used to perform extra-oral antisepsis. The surgical site was anaesthetized. A mucoperiosteal flap was elevated and reflected followed by thorough debridement of all inflammatory granulation tissue from IBD until a sound, healthy bone surface was obtained. Root surface debridement was also performed. Copious irrigation with normal saline solution. A mixture of Ly-PRF and n-HA (1:1by weight) was hydrated with a few drops of normal saline then, it was applied and packed to fill the defect. The flap was repositioned and sutured.
  Interventions: Biological: open flap debridement

INTERVENTIONS:
Biological: open flap debridement — does lyophilized platelet rich fibrin combined with open flap debridement or combination of open flap debridement, lyophilized platelet rich fibrin and nano-crystalline hydroxyapatite bone substitute can add benefits to open flap debridement alone or not
  Other Names: lyophilized platelet rich fibrin combined with open flap debridement; combination of lyophilized platelet rich fibrin and nano-crystalline hydroxyapatite bone substitute

SUMMARY:
The present study will be performed to evaluate the efficacy of lyophilized platelet-rich fibrin alone and combined with nanocrystalline hydroxyapatite in treatment of periodontal intra-bony defects through:

1. Primary outcomes:

   * The clinical parameters including: Probing pocket depth (PPD) reduction and clinical attachment level (CAL) gain.
   * The radiographic parameters including: Marginal bone level (MBL), bone-defect fill.
2. Secondary outcome: The level of BMP-2 in Gingival crevicular fluid (GCF).

DETAILED DESCRIPTION:
Periodontitis is a multi-factorial inflammatory process affecting the periodontal tissues. Among the characteristic signs of periodontal disease is loss of alveolar bone support. The risk of further alveolar bone loss and the probability of tooth loss increases with the presence of intra-bony defects.

Periodontal intra-bony defects (IBDs) are osseous defects with specific morphology, the bottom of these defects is located more apically than the alveolar crest and they are surrounded by bony walls on 1-, 2-, or 3- sides, with the tooth root forming the additional wall. The prevalence of these defects is significantly lower than supra-crestal periodontal defects.

Among the main goals of periodontal therapy is to regenerate the lost periodontal tissues after arresting the progress of the disease. Surgical management of periodontally affected sites includes conventional and regenerative procedures. The conventional modality of surgical debridement allows for reliable access to root surfaces leading only to healing by repair. While the regenerative treatment options allow for the regeneration of destroyed periodontal ligament and bone. Guided tissue regeneration (GTR), placement of bone grafting materials, the addition of biologic mediators and a combination of such techniques are the different forms of periodontal regenerative techniques.

Bone grafts (BGs) and substitutes are classified into autogenic, allogenic, xenogenic and synthetic bone grafts. Synthetic nanocrystalline hydroxyapatite (NCHA) has been extensively applied as bone graft replacement material and characterized by its osteoconductive properties and improved osseointegrative features. The size of the particle was found to be around 18 nm, allowing for quicker vital bone substitution. It has been proved that NCHA can enhance the adhesion of the bone formative cells (osteoblasts) more than micromaterials. Furthermore, the nano-sized particles provide special properties to NCHA such as ahydrated surface layer, a large surface/volume ratio, this layer is actively involved in the homeostasis process, ionic exchange and other techniques involved in the osteogenesis regulation. NCHA is osteoconductive but has inferior osteoinductive properties; therefore, one of the efforts to increase the ability of this material is to combine it with other bioactive materials such as platelet-rich fibrin (PRF).

Platelet-rich fibrin is a second-generation platelet concentrate that has been widely used in the treatment of bone deficiency and its main action is derived from its high content of platelets that release many growth factors (GFs) and cytokines. However, freshly prepared PRF must be used immediately in order to retain the bioactivity of growth factors. In addition, the bio-degradation rate of PRF is fast and irregular, along with the rapid release of growth factors, and then enzymatically hydrolyzed.

The lyophilization of PRF by vacuum freeze dryer was found to provide a dense three-dimensional fibrin network, better storage stability with a longer half-life and preservation of GFs. Lyophilized platelet-rich fibrin (Ly-PRF) showed adaptability as a viable biomaterial for application as a craniofacial bio-scaffold due to, the advantage of lowering the difficulty in application, providing a newly grown tissue with straightforward access to multiple GFs as well as, sustained release GFs presenting a better tissue regeneration process and bone tissue reconstruction.

It was proven that, Ly-PRF significantly improve the osteogenic differentiation of bone marrow mesenchymal stem cell (BMSC) in vitro through the upregulation of osteogenic markers: collagen type I, osteopontin (OPN), osteocalcin (OCN), and bone morphogenetic protein 2 (BMP-2). BMP-2 is described as being osteoinductive, which is capable of inducing and enhancing bone growth and formation, and it also promotes cell chemotaxis, proliferation and differentiation towards the osteogenic pathway.

The present clinical trial will be performed to clarify and shed some light on Ly-PRF in periodontal regeneration

ELIGIBILITY:
Inclusion Criteria:

* All periodontitis patients to be included in this study should be diagnosed as having stage III periodontitis with probing pocket depth (PPD) ≥ 6 mm, and clinical attachment loss (CAL) ≥ 5mm.
* 2- or 3-wall intra-bony interproximal defect with depth ≥3 mm, a width of ≥3 mm at its most coronal part and 45-55-degree angulation will be selected in order to reduce defect variability.
* All patients will be free from any systemic diseases according to the American Dental Academy general guidelines for referring dental patients to specialists and other care settings

Exclusion Criteria:

* Any patients with any systemic condition that contraindicate any surgical intervention.
* Pregnant or lactating females, smokers, or alcoholic patients.
* Patients with intra-bony defects received drugs that affect bone turnover such as (chemotherapy and radiotherapy).
* History of periodontal therapy and antibiotic administration in the last 6 months.
* Patients taking any medicine which may affect the function of platelet (i.e., aspirin) in the previous 3 months.
* Miller grade II or greater mobility, furcation involvement as well as one-wall defects and interdental craters.
* Patients with unacceptable oral hygiene after the re-evaluation of phase I therapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
radiographic parameters | baseline, 3, 6, and 9 months after treatment
  The radiographic parameters including: Bone-defect fill in mm.
clinical parameters | baseline, 3, 6, and 9 months after treatment.
  The clinical parameters including: Clinical attachment level (CAL) gain in mm.

SECONDARY OUTCOMES:
biochemical evaluation | baseline, 1, 4 and 12 weeks after surgery
  The level of BMP-2 (Pg/ml) in Gingival crevicular fluid (GCF).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Al- Azhar University,, Asyut, Egypt

REFERENCES:
- [Background] Anoixiadou S, Parashis A, Vouros I. Minimally Invasive Non-Surgical Technique in the Treatment of Intrabony Defects-A Narrative Review. Dent J (Basel). 2023 Jan 11;11(1):25. doi: 10.3390/dj11010025. PMID 36661562
- [Background] Tavelli L, Chen CJ, Barootchi S, Kim DM. Efficacy of biologics for the treatment of periodontal infrabony defects: An American Academy of Periodontology best evidence systematic review and network meta-analysis. J Periodontol. 2022 Dec;93(12):1803-1826. doi: 10.1002/JPER.22-0120. Epub 2022 Oct 24. PMID 36279121
- [Background] Zhao R, Yang R, Cooper PR, Khurshid Z, Shavandi A, Ratnayake J. Bone Grafts and Substitutes in Dentistry: A Review of Current Trends and Developments. Molecules. 2021 May 18;26(10):3007. doi: 10.3390/molecules26103007. PMID 34070157
- [Background] Shaikh MS, Zafar MS, Alnazzawi A, Javed F. Nanocrystalline hydroxyapatite in regeneration of periodontal intrabony defects: A systematic review and meta-analysis. Ann Anat. 2022 Feb;240:151877. doi: 10.1016/j.aanat.2021.151877. Epub 2021 Dec 2. PMID 34864225
- [Background] Liu X, Yin M, Li Y, Wang J, Da J, Liu Z, Zhang K, Liu L, Zhang W, Wang P, Jin H, Zhang B. Genipin modified lyophilized platelet-rich fibrin scaffold for sustained release of growth factors to promote bone regeneration. Front Physiol. 2022 Sep 30;13:1007692. doi: 10.3389/fphys.2022.1007692. eCollection 2022. PMID 36246111
- [Background] Wang Z, Han L, Sun T, Wang W, Li X, Wu B. Preparation and effect of lyophilized platelet-rich fibrin on the osteogenic potential of bone marrow mesenchymal stem cells in vitro and in vivo. Heliyon. 2019 Nov 1;5(10):e02739. doi: 10.1016/j.heliyon.2019.e02739. eCollection 2019 Oct. PMID 31720476
- [Background] Ngah NA, Dias GJ, Tong DC, Mohd Noor SNF, Ratnayake J, Cooper PR, Hussaini HM. Lyophilised Platelet-Rich Fibrin: Physical and Biological Characterisation. Molecules. 2021 Nov 25;26(23):7131. doi: 10.3390/molecules26237131. PMID 34885714
- [Background] Zhu L, Liu Y, Wang A, Zhu Z, Li Y, Zhu C, Che Z, Liu T, Liu H, Huang L. Application of BMP in Bone Tissue Engineering. Front Bioeng Biotechnol. 2022 Mar 31;10:810880. doi: 10.3389/fbioe.2022.810880. eCollection 2022. PMID 35433652
- [Result] Tsoromokos N, Parinussa S, Claessen F, Moin DA, Loos BG. Estimation of Alveolar Bone Loss in Periodontitis Using Machine Learning. Int Dent J. 2022 Oct;72(5):621-627. doi: 10.1016/j.identj.2022.02.009. Epub 2022 May 13. PMID 35570013
- See also: Combination of Nanocrystalline Hydroxyapatite and Injectable Platelet-Rich Fibrin on Bone Graft Materials for Alveolar Bone Preservation — https://oamjms.eu/index.php/mjms/article/view/8762